CLINICAL TRIAL: NCT04813159
Title: Remote Ischaemic Conditioning in STEMI Patients in AFRICA: The RIC-AFRICA Trial
Brief Title: Remote Ischaemic Conditioning in STEMI Patients in AFRICA
Acronym: RIC-AFRICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Groote Schuur Hospital, South Africa (Unknown); Uganda Heart Institute (Other); Mombasa Hospital, Kenya (Unknown); Coast General Teaching Hospital, Kenya (Unknown); Kenyatta National Hospital (Other Government); Al Shaab Teaching Hospital, Sudan (Unknown); Sudan Heart Centre, Sudan (Unknown); Aliaa Specialist Hospital, Sudan (Unknown); Medani Heart Centre, Sudan (Unknown); Al Saha Specialised Hospital, Sudan (Unknown); Omdurman Hospital, Sudan (Unknown); Victoria Hospital, South Africa (Unknown); George Hospital, South Africa (Unknown); Charlotte Maxeke Hospital, South Africa (Unknown); Tshepong Hospital, South Africa (Unknown); Wentworth Hospital, South Africa (Unknown); Grey's Hospital (Other); Universitas Academic Hospital, South Africa (Unknown); University College, London (Other); Royal Care international Hospital, Sudan (Unknown); Nairobi West Hospital, Kenya (Unknown)
Responsible Party: Principal Investigator, Mpiko Ntsekhe, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIC AFRICA
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-12

CONDITIONS: STEMI; Remote Ischaemic Conditioning; Myocardial Reperfusion Injury
Keywords: Cardioprotection; Ischaemia/reperfusion injury; ST-Elevation myocardial infarction; Hospitalisation for post-myocardial infarction heart failure; Remote Ischaemic Conditioning; Cardiovascular mortality; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Reperfusion Injury; Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: Consented participants presenting with STEMI within 24 hours and who fulfil the study's eligibility criteria will be assigned a participant identification number and randomised to receive either RIC or sham control in a 1:1 ratio to ensure equal distribution amongst experimental arm. Randomisation will be conducted via a secure website and will be stratified by recruiting centre and patient stratum to ensure that a minimum of 2 participants in stratum 1 (eligible for thrombolysis and within <12 hours of MI onset) are recruited for every participant in stratum 2 (ineligible for thrombolysis because they present outside of guideline-recommended time (<12 hours) but presenting within 24 hours of most severe chest pain onset). The patient, treating clinician, study investigator and research team analysing the data will be blinded to the treatment allocation. Study intervention will be applied by the research nurse who will not have any further contact with the participant or trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, treating clinician, study investigator and research team analysing the data will be blinded to the treatment allocation. Study intervention will be applied by the research nurse who will not have any further contact with the participant or trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Remote Ischaemic Conditioning (RIC) (Active Comparator): Consented STEMI participants presenting < 24 hours who are randomised to the RIC protocol, will receive blood pressure cuff inflation by the automated RIC blood pressure device to 20 mmHg above systolic blood pressure for 5 minutes and deflation for a further 5 minutes, a cycle which will be completed four times in total. The RIC protocol will be repeated daily for the next 2 days.
  Interventions: Device: Remote Ischaemic Conditioning (RIC)
- Sham-control (Sham Comparator): Consented STEMI participants presenting < 24 hours who are randomised to the sham protocol will receive low-pressure cuff inflation to 20 mmHg for 5 minutes and deflation for a further 5 minutes, a cycle which will be completed four times in total by a visually identical pneumatic cuff. The sham control protocol will be repeated daily for the next 2 days.
  Interventions: Device: Sham-control
- Observational (No Intervention): Consented STEMI participants presenting > 24 hours but within 72 hours of MI onset will be recruited into the observational arm of the study which will have the same study endpoints as the RCT. These participants will not be randomised or receive any trial intervention.

INTERVENTIONS:
Device: Remote Ischaemic Conditioning (RIC) — The RIC protocol will comprise inflation of the automated RIC device to 20 mmHg above systolic blood pressure for 5 minutes and deflation for a further 5 minutes, a cycle which will be completed four times in total. The RIC protocol will be repeated daily for the next 2 days.
  Arms: Remote Ischaemic Conditioning (RIC)
Device: Sham-control — The sham protocol will comprise low-pressure inflation to 20 mmHg for 5 minutes and deflation for a further 5 minutes, a cycle which will be completed four times in total by a visually identical pneumatic cuff used in the active arm. The sham control protocol will be repeated daily for the next 2 days.
  Arms: Sham-control

SUMMARY:
The RIC-AFRICA trial is a multi-centre, sham-controlled, randomised controlled trial (RCT) involving 1400 ST-segment elevation myocardial infarction (STEMI) patients presenting within ≤ 24 hours of myocardial infarction (MI) onset, across approximately 25 sites in 7 African countries (South Africa, Kenya, Sudan, Uganda, Mozambique, Senegal and Mauritius). Patients presenting with STEMI and deemed ineligible for the RIC AFRICA RCT because they present >24 hours from MI onset but less than 72 hours, will be recruited into the observational arm of the study with the same endpoints as the trial. The purpose of the RCT is to determine whether Remote Ischaemic Conditioning (RIC) can reduce the rates of all-cause death and early post-myocardial heart failure at 30-days in STEMI patients treated predominantly with thrombolytic therapy.

DETAILED DESCRIPTION:
Background:

Remote ischaemic conditioning (RIC) using transient limb ischaemia and reperfusion has been shown to reduce myocardial infarct size in animal studies and small proof-of-concept clinical studies in ST-segment elevation myocardial infarction (STEMI) patients. However, RIC failed to improve clinical outcomes in the large European CONDI-2/ERIC-PPCI multi-centre randomised clinical trial. Potential reasons for this failure include the low-risk patients recruited into the study and the fact that patients received timely and optimal reperfusion therapy by primary percutaneous coronary intervention. The RIC-AFRICA trial will investigate whether RIC can improve clinical outcomes in higher-risk STEMI patients treated by thrombolysis in Africa.

Study design:

The RIC-AFRICA trial is a multi-centre, sham-controlled, randomised controlled trial (RCT) involving 1400 ST-segment elevation myocardial infarction (STEMI) patients presenting within ≤ 24 hours of myocardial infarction (MI) onset, across approximately 20 sites in 7 African countries (South Africa, Kenya, Sudan, Uganda, Mozambique, Senegal and Mauritius). Patients will be randomised to receive either RIC or sham control initiated prior to thrombolysis and applied daily for the next 2 days. The RIC protocol will comprise four 5-minute cycles of inflation (to 20mmHg above systolic blood pressure) and deflation of an automated pneumatic cuff placed on the upper arm. The sham control protocol will comprise four 5-minute cycles of low-pressure inflation (to 20mmHg) and deflation by a visually identical pneumatic cuff. The primary composite endpoint will be all-cause death and new-onset heart failure at 30-days post STEMI. Patients presenting with STEMI and deemed ineligible for the RIC AFRICA RCT because they present >24 hours from MI onset but less than 72 hours, will be recruited into the observational arm of the study with the same endpoints as the trial.

Implications:

The RIC-AFRICA trial will determine whether RIC can reduce rates of death and prevent heart failure in higher-risk STEMI patients treated by thrombolytic therapy in Africa, thereby potentially providing a low-cost, non-invasive therapy for improving health outcomes.

ELIGIBILITY:
We will be recruiting 3 different strata of STEMI patients.

1. Adult patients (≥18 years old) presenting with STEMI receiving thrombolytic therapy within guideline-recommended time (i.e., within <12 hours of most severe chest pain onset).
2. Adult patients (≥18 years old) presenting with STEMI who are ineligible for thrombolysis because they present outside of guideline-recommended time (<12 hours) but within 24 hours of most severe chest pain onset.
3. Adult patients (≥18 years old) presenting with evidence of STEMI who do not receive thrombolysis and who present ≥24 hours and within 72 hours of most severe chest pain onset.

Interventional arm of the Study: Randomized Control Trial

Patients who are deemed eligible for randomization into the trial on account of presentation with STEMI within 24 hours, will be eligible for the interventional arm of the study if the following inclusion/exclusion criteria are met.

Inclusion Criteria

I. Adult patients (≥18 years old) presenting with suspected STEMI (ST-elevation at the J-point in two contiguous leads ( ≥ 0.2mV in men or ≥ 0.15mV in women in leads V2-V3 and/or ≥ 0.1mV in other lead); and II. Within 24 hours of onset of myocardial infarction as deemed by the attending clinician; and III. Signed informed consent.

Exclusion criteria

I. STEMI patients due to undergo primary percutaneous coronary intervention;

II. STEMI patients presenting with cardiogenic shock or haemodynamic instability as defined by: systolic blood pressure (SBP) measurement of <90 mm Hg for ≥30 minutes; or use of pharmacological and/or mechanical support to maintain SBP ≥ 90 mm Hg; and evidence of end-organ damage defined by: urine output of <30 mL/h; altered mental status; and/or serum lactate >2.0 mmol/L;

III. Contraindications for the use of RIC or sham-control on either arm such as:

1. severe active skin disease/burns on both arms; or
2. bilateral upper limb amputations; or
3. evidence of acute limb ischaemia on either arm; or
4. active upper limb gangrene of any digits;
5. breast cancer with lymph-node involvement on the ipsilateral side of RIC; or
6. bilateral arteriovenous fistulae needed for haemodialysis.

IV. Inter-current disease with an expected life expectancy of less than 24 hours;

V. Contra-indication to thrombolytic therapy in patients presenting within guideline-recommended time (<12 hours).

Observational arm of the study

Patients who are deemed ineligible for randomization into the trial on account of presentation beyond 24 hours, will be eligible for the observational arm of the study if the following inclusion/exclusion criteria are met.

Inclusion Criteria

I. Signed informed consent; and

II. Clinical evidence of STEMI older than 24 hours and less than 72 hours as defined by:

1. Compatible history with maximal chest pain between 24 -72 hours prior to presentation; and
2. Compatible biomarkers (elevated cardiac troponin); and
3. ECG compatible with recent STEMI; and/or
4. Compatible echocardiography.

Exclusion criteria

I. Refusal or inability to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death and early post-MI heart failure | 30 days
  The primary endpoint of the study will be a composite of all-cause death and early post-MI heart failure. The latter describes both a] pre-discharge (in-hospital) heart failure; or b] post discharge heart failure hospitalisation within 30 days for patients discharged free of heart failure after the index MI admission.

SECONDARY OUTCOMES:
Composite clinical endpoint for MACCE | 30 days
  Secondary outcome measures will include a composite clinical endpoint of MACCE at 30 days follow-up, defined as rates of (i) all-cause mortality; (ii) non-fatal myocardial infarction; (iii) transient ischaemic attack or stroke; and (iv) heart failure with or without hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Mpiko Ntsekhe, PhD, Principal Investigator — University of Cape Town; Derek Hausenloy, PhD, Principal Investigator — Hatter Cardiovascular Institute; Derek Yellon, PhD, Principal Investigator — Hatter Cardiovascular Institute; Malcolm Walker, PhD, Principal Investigator — Hatter Cardiovascular Institute
Locations (20):
- Kenya (4):
  - Coast General Teaching Hospital, Mombasa, Mombasa County
  - Mombasa Hospital, Mombasa, Mombasa County
  - Kenyatta National Hospital, Nairobi, Nairobi County
  - Nairobi West hospital, Nairobi
- Hospital Central de Mpauto, Maputo, Mozambique
- Hopital Principal de Dakar, Dakar, Senegal
- South Africa (7):
  - Charlotte Maxeke Hospital, Johannesburg, Gauteng
  - Wentworth Hospital, Durban, KwaZulu-Natal
  - Tshepong Hospital, Klerksdorp, North West
  - Mitchell's Plain District Hospital, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Victoria Hospital, Cape Town, Western Cape
  - George Hospital, George, Western Cape
- Sudan (6):
  - Al Saha Specialised Hospital, Khartoum, Khartoum State
  - Al Shaab Teaching Hospital, Khartoum, Khartoum State
  - Sudan Heart Centre, Khartoum, Khartoum State
  - The Royal Care International Hospital, Khartoum, Khartoum State
  - Aliaa Specialist Hospital, Omdurman, Omdurman
  - Medani Heart Centre, Wad Medani
- Uganda Heart Institute, Kampala, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lukhna K, Hausenloy DJ, Ali AS, Bajaber A, Calver A, Mutyaba A, Mohamed AA, Kiggundu B, Chishala C, Variava E, Elmakki EA, Ogola E, Hamid E, Okello E, Gaafar I, Mwazo K, Makotoko M, Naidoo M, Abdelhameed ME, Badri M, van der Schyff N, Abozaid O, Xafis P, Giesz S, Gould T, Welgemoed W, Walker M, Ntsekhe M, Yellon DM. Remote Ischaemic Conditioning in STEMI Patients in Sub-Saharan AFRICA: Rationale and Study Design for the RIC-AFRICA Trial. Cardiovasc Drugs Ther. 2023 Apr;37(2):299-305. doi: 10.1007/s10557-021-07283-y. Epub 2021 Nov 5. PMID 34739648